CLINICAL TRIAL: NCT07052045
Title: One-Stop manaGemEnT For A Swift Initiation of Endovascular Therapy - An International, Multicenter, Pragmatic Randomized Controlled Trial (GET-FAST
Brief Title: One-Stop manaGemEnT For A Swift Initiation of Endovascular Therapy
Acronym: GET-FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Jan Liman (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Deutsche Forschungegemeinschaft (Unknown); Klinikum Nürnberg (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jan Liman, Prof. Dr., Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GET-FAST
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke Acute; Acute Ischemic Stroke AIS; Hemorrhagic Stroke, Intracerebral
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One Stop Management (Experimental): Patients within the intervention group will be transported directly after randomization to the angiography room.
  Interventions: Other: One Stop Management
- Usual Care Management (Active Comparator): Patients within the control group will be transported directly after randomization to the multidetector CT (MDCT) room for diagnostic imaging with non-contrast MDCT and MDCT-A.
  Interventions: Other: Usual care management

INTERVENTIONS:
Other: One Stop Management — Patients within the intervention group will be transported directly after randomization to the angiography room. In the angiography room diagnostic imaging will be performed using cranial non-contrast FDCT and FDCT-A with subsequent EVT (if a treatable vessel occlusion was identified). Therefore, diagnostics and treatment will be performed in the same room (One-Stop management). Only patients with a treatable occlusion will undergo arterial puncture.
  Arms: One Stop Management
Other: Usual care management — Patients within the control group will be transported directly after randomization to the multidetector CT (MDCT) room for diagnostic imaging with non-contrast MDCT and MDCT-A. IVT will be given directly in the MDCT room if no contraindication is present. If on diagnostic imaging a treatable vessel occlusion was identified, the patient will be transported to the angiography room, where EVT will be performed.
  Arms: Usual Care Management

SUMMARY:
Stroke, especially acute ischemic stroke (AIS) caused by a blocked blood vessel in the brain, is a leading cause of death and long-term disability. When the blockage is in a large blood vessel, a procedure called endovascular therapy (EVT)-where the clot is removed using a catheter-is highly effective. However, the sooner EVT is done, the better the outcome for the patient.

Research has shown that delays between arriving at the hospital and starting EVT (called door-to-groin time) significantly reduce the chances of recovery. For example, reducing this time by just 15 minutes can mean 20 more patients (out of 1,000 treated) going home instead of to a care facility. Even a 10-minute improvement can result in over 100 extra days of independent living for patients and save more than $10,000 in healthcare costs per patient.

To reduce these delays, hospitals have improved stroke workflows. In the current standard approach, patients suspected of having a stroke are taken first to a CT scan room to confirm the diagnosis, and then, if a treatable occlusion is found, to a separate room for EVT. This usually takes around 60-70 minutes.

However, moving patients between rooms takes time. A new approach called "One-Stop management" could solve this. In this method, both the brain scan and the EVT procedure are done in one room-the angiography suite-using special imaging tools called flat panel CT (FDCT) and FDCT angiography (FDCT-A).

A previous study with 230 patients showed that One-Stop management is possible and saves time. But there's a challenge: the decision to follow the One-Stop pathway is made before a clear diagnosis is available. That's important because not all strokes benefit from EVT. Severe stroke symptoms (measured by a score called NIHSS ≥10) can come from:

* A large or medium vessel blockage (which EVT can treat),
* A small vessel blockage, or
* A bleed in the brain (hemorrhage). Only the first group benefits from EVT. About 85% of patients with severe symptoms fall into this category. The rest-about 15%-would not benefit, and there are concerns that FDCT might be slightly less accurate than regular CT in diagnosing these types of strokes. So, we need to test whether One-Stop management is safe and effective for all patients, not just those with treatable blockages.

To do this, the GET-FAST trial will compare the One-Stop approach to the standard two-room process. Patients will be randomly assigned to one of the two strategies. Importantly, this randomization won't affect their actual treatment-everyone will still receive the best care according to current medical guidelines. The main endpoint for the evaluation of the One-Stop approach will be long-term (at 90 days) disability and dependency in daily life as measured with the modified Rankin Scale (mRS).

This study will include all patients as they were assigned, regardless of what type of stroke they actually had. This is called an "intention-to-treat" analysis, and it provides the most reliable measure of the overall impact of One-Stop management.

Another key aspect of the trial is that any CE-certified imaging system already used in hospitals can be used for the One-Stop process-no specific brand or model is required. This makes the results more applicable to real-world hospital settings.

If GET-FAST proves that One-Stop management leads to better patient outcomes, this could transform how stroke care is delivered. More patients could return to independent living, and fewer would require long-term care -leading to major reductions in healthcare costs. For example, even a one-point improvement on a common stroke disability scale (mRS) can triple the savings in lifetime care costs.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suggestive of an acute ischemic stroke caused by a large or medium vessel occlusion as defined by a National Institute of Health Stroke Scale (NIHSS) Score of ≥ 10 points
* Patient presents directly to the treating hospital (mothership patient) within 4.5 hours of last seen well (LSW)
* Age ≥ 18 years
* Patient was independent in daily activities prior to the stroke (pre stroke modified Rankin Scale of 0 - 2)
* Endovascular treatment team available (Neurologist, Interventionist, Anesthesiologist, Nursery, Technicians)
* Informed Consent as documented by signature or fulfilling the criteria for emergency consent procedures

Exclusion Criteria:

* Severe comorbidities, which will likely prevent improvement or follow-up
* In-hospital stroke
* Clinical symptoms suggestive of intracranial hemorrhage (deterioration of patient during transport, vomiting or depressed consciousness)
* Strong suspicion of functional neurological symptom disorder / conversion disorder
* Hemodynamically unstable patients who require advanced vital support
* Angiography room occupied by other procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Degree of Dependency and disability in daily activities | 90 days (+/- 15 days) after randomization
  As assessed with the modified Rankin Scale (mRS); The mRS runs from 0-6, running from perfect health without symptoms (0) to death (6).

SECONDARY OUTCOMES:
Early neurological improvement | 5 - 7 days after randomization or discharge if earlier
  Early neurological improvement is defined as a decrease of at least 4 points on the National Institute of Health Stoke Scale (NIHSS) compared to baseline; range of NIHSS 0 - 42 with higher values indicating more severe neurological deficit
Early neurological deterioration | 5 - 7 days after randomization or discharge if earlier
  Early neurological deterioration is defined as an increase of at least 4 points on National Institutes of Health Stroke Scale compared to baseline, death or persistent coma; range of NIHSS 0 - 42 with higher values indicating more severe neurological deficit
Independent functional outcome | 90 days (+ / - 15 days) after randomization
  Defined as a modified Rankin Scale of 0 to 2 (mRS); The mRS runs from 0-6, running from perfect health without symptoms (0) to death (6).
Cognitive function | 90 days (+/- 15 days) after randomization
  As assessed with the Montreal Cognitive Assessment Test (MoCA); range 0 - 30 with lower values indicating more severe cognitive impairment
Health-related quality of life | 90 days (+/- 15 days) after randomization
  As assessed with the Euro-Qol 5d; 5 point scale with higher values indicating better quality of life in the specific domain
Degree of Dependency and disability in daily activities | 365 days (+/- 30 days) after randomization
  As assessed with the modified Rankin Scale (mRS); The mRS runs from 0-6, running from perfect health without symptoms (0) to death (6).
Health-related quality of life | 365 days (+/- 30 days) after randomization
  As assessed with the Euro-QoL-5D; 5 point scale with higher values indicating better quality of life in the specific domain
Cognitive function | 365 days (+/- 30 days) after randomization
  As assessed with the telephone Montreal Cognitive Assessment Test (T-MoCA); range 0 - 22 with lower values indicating more severe cognitive impairment

OTHER OUTCOMES:
Safety: Symptomatic intracranial hemorrhage | Within 24 hours (+/- 12 hours) after randomization
  All intracerebral hemorrhages will be classified by the blinded Core Lab according to the Heidelberg Bleeding Classification.
  Symptomatic intracerebral hemorrhage (sICH) will be defined using a modified SITS-MOST definition:
  sICH is defined as the presence of a parenchymal hemorrhage type 2 (local or remote), subarachnoid hemorrhage, and/or intraventricular hemorrhage on imaging performed 24 hours post-treatment (±12 hours), in combination with one of the following: A neurological deterioration of ≥4 points on the National Institute of Health Stroke Scale (NIHSS; ranging from 0 - 42 with higher values indication more severe neurological deficit) from baseline, or from the lowest NIHSS value between baseline and 24 hours; persistent coma; or Death.
Safety: Serious Adverse Events | Within 90 days after randomization
Safety: Mortality | Within 90 days after randomization
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jan Liman, Dr, Principal Investigator — Klinkum Nuremberg; Marios Psychogios, Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Klinik für Neurologie, Universitätsklinik der Paracelsus, Nuremberg, Germany
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 years after publication of the main results with no end date.
Access Criteria: A proposal that describes the planned analyses shall be submitted to the sponsor-investigator of the trial.

REFERENCES:
- [Background] Psychogios MN, Behme D, Schregel K, Tsogkas I, Maier IL, Leyhe JR, Zapf A, Tran J, Bahr M, Liman J, Knauth M. One-Stop Management of Acute Stroke Patients: Minimizing Door-to-Reperfusion Times. Stroke. 2017 Nov;48(11):3152-3155. doi: 10.1161/STROKEAHA.117.018077. Epub 2017 Oct 10. PMID 29018132
- [Background] Psychogios MN, Maier IL, Tsogkas I, Hesse AC, Brehm A, Behme D, Schnieder M, Schregel K, Papageorgiou I, Liebeskind DS, Goyal M, Bahr M, Knauth M, Liman J. One-Stop Management of 230 Consecutive Acute Stroke Patients: Report of Procedural Times and Clinical Outcome. J Clin Med. 2019 Dec 11;8(12):2185. doi: 10.3390/jcm8122185. PMID 31835763
- See also: Related Info — https://onestopinstroke.eu